CLINICAL TRIAL: NCT05374434
Title: Comparative Evaluation of the Effectiveness of Root Canal Preparation After Irrigation Using Endodontic Needle and Inertial Cavitation: A Randomized Controlled Trial
Brief Title: A First in Human Study to Compare Feasibility of Inertial Cavitation Irrigation to SNI in Root Canal Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumendo AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: LUM-EC-001-060522
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Root Canal Treatment; Post Operative Pain
Keywords: Root Canal Irrigation; Root Canal Cleaning; Root Canal Treatment; Post Operative Pain; Root Canal Disinfection; Inertial cavitation; NaOCl Irrigation; Debridement
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional irrigation (Active Comparator): Root canal cleaning will be performed by manual irrigation with sodium hypochlorite NaOCl solution.
  Interventions: Other: Conventional irrigation
- Inertial cavitation (Experimental): Root canal cleaning will be performed by inertial cavitation-generating device.
  Interventions: Device: Inertial cavitation

INTERVENTIONS:
Other: Conventional irrigation — The participant will be treated by manual irrigation with sodium hypochlorite NaOCl.
  Arms: Conventional irrigation
Device: Inertial cavitation — The participant will be treated by inertial cavitation-generating device, that generates hydraulic cavitation to clean root canals deeper and more effectively than other existing systems.
  Arms: Inertial cavitation

SUMMARY:
The study design is a single-center 2-arm randomized controlled clinical trial. 10 subjects (teeth) requiring a root canal treatment will be enrolled in 2 groups (5 in each group). The aim of the study is to compare the postoperative pain intensity levels in patients with asymptomatic teeth diagnosed for non-surgical orthograde root canal treatment that are disinfected during the root canal treatment procedure by manual irrigation with sodium hypochlorite (NaOCl) solution using an endodontic needle or by a inertial cavitation-generating device.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Physical status classification system described was used for patients' recruitment. Healthy patients, who were classified by the American Society of Anaesthesiologists (ASA) as ASA I and II
2. Patients with the age of 18 and over
3. Patients who were diagnosed as in need of non-surgical orthograde root canal treatment of an asymptomatic tooth
4. Tooth without signs of previously initiated Root Canal Therapy

Exclusion Criteria:

1. Pregnant and lactating females
2. Patients with chronic periodontal diseases
3. Patients with sensitivity or adverse reactions to any medication or materials that were used throughout the treatment procedure
4. Patients with acute periapical periodontitis
5. Patients with acute periodontal abscess
6. Patients who could not abide by the follow-up time
7. Patients who used analgesics 1-week prior or antibiotics 1-month prior to treatment
8. Uncooperative patients
9. Teeth that cannot be made functional nor restored or difficult to access teeth with no importance (wisdom teeth)
10. Teeth with poor prognosis, for example, due to deep root caries or big root resorption
11. Teeth with 4 mm periodontal pocket depth
12. Teeth with an inaccessible root end
13. Teeth with apical resorption or a radiologically not clearly defined apex
14. Fractured teeth
15. Teeth with immature or open apices Confidential
16. Teeth with root apices extending into the maxillary sinus

All treatment procedures will be performed in a single visit by a single treatment provider. It will be assured that the operation room is quiet and isolated throughout the whole process to avoid any outside interference. Patients will be made comfortable and informed about the steps of the procedure a second time right before commencing the treatment protocol. Patients will be also reminded that they will get the necessary treatment even if they decline from the study and should not feel compelled to participate the study for a proper treatment. All root canal treatments will be performed using a dental loupe with a magnification of 4.50X (EyeMag Pro F; Carl Zeiss).

Each tooth will be anaesthetized with 2 mL local anaesthetic solution containing 40 mg/mL articaine hydrochloride and 12 mg/mL epinephrine hydrochloride (Ultracaine DS Forte; Aventis Pharma). After isolating the tooth with a rubber dam (Hygenic Dental Dam Kit; Coltene/Whaledent Gmbh & Co.kg, Langenau, Germany) the operation field will be disinfected using 5.25% NaOCl solution (Wizard; Rehber Chemistry) soaked cotton rolls. After the access cavity preparation, a #10 C-File (MMC file, Coltene-Micro-Méga, Besançon, France) will be introduced into the root canal for scouting. Coronal flaring of root canals will be performed using a nickel-titanium flaring file (One Flare; Coltene-Micro-Méga) with an electric endodontic motor (Dual Move, Coltene-Micromega). Working length determination will be performed with a #10 C-file (MMC file, Coltene-Micro-Méga) and glidepath preparation will be completed with a One G (Coltene-Micro-Méga). The shaping of the root canals will be performed using One Curve (#25/0.06, Coltene-Micro-Méga). If further shaping of the canal will be needed 2 Shape F35 (#35/0.06) (ColteneMicro-Méga) files will be used according to apical canal lumen. All rotary files will be used according to the manufacturer's instructions. The filing protocols and files used will be recorded in the patient file.

In Group 1, 2 mL of NaOCl solution will be used after each file as an irrigation solution. After the shaping of the root canal is completed final irrigation with a 31G double side vented tip is performed in each canal using 2.5 mL of 5% EDTA (Wizard; Rehber Chemistry) for 1 minute, 2.5 mL of 5.25% NaOCl for 30 seconds and 5 mL of saline solution for 30 seconds respectively.

In Group 2, 2 mL of NaOCl solution will be used after each file as an irrigation solution. After the shaping of the root canal is completed, the NaOCl solution is removed from the root canal with 2.5 mL saline solution using a syringe with a 31G needle. EndoClean tip is introduced into the root canal, always maintaining a distance of at least 3mm from the apex. The EndoClean device is used for 60 seconds for each root canal.

In both groups, following root canal preparation, a matching gutta-percha cone (#25/0.06 or #35/0.06) (MM GP Points, Coltene-Micro-Méga) is introduced into the root canal coated with a calcium silicate-based root canal sealer (BioRoot RCS; Lancester PA, USA). Single-cone technique is used to fill the root canals.

Total-etch technique is used to restore the coronal part of each tooth. The cavities are etched with 35% H3PO4 for 15 seconds before a single layer application of an adhesive material (Adper Single Bond 2; 3M ESPE). After photopolymerization (Elipar S10, 3M ESPE) of the adhesive material for 20 seconds, a flowable bulk-fill composite material (Estelite, BulkFill Flow, Tokuyama Dental, Tokyo, Japan) is used to restore the coronal cavity incrementally with a thickness of 4 mm for every layer. Each layer is photopolymerized for 20 seconds.

Post-endodontic pain assessment :

After the treatment, all participants will be provided with analgesics (75 mg diclofenac sodium) (Voltaren SR 75 mg, Novartis, Kurtköy, İstanbul) and will be advised to use them if needs be and record the time of use. A pain intensity evaluation diary including VAS diagrams with their respective follow-up evaluation times will be provided to each participant to mark their pain. All participants will be contacted on their follow-up time to remind them to mark their pain intensity scores. Pain intensity of patients will be evaluated at 6h, 24h, 48h, 72h and 1 week after the completion of root canal treatment as previously described. Any complication such as paraesthesia, acute exacerbations, flare-ups, swellings will be also recorded on patients' charts. Patients who fail to abide by the followup time will be traced via phone, e-mail or SMS to determine the possible reasons for dropout.

ELIGIBILITY:
Inclusion Criteria:

1. Physical status classification system described was used for patients' recruitment. Healthy patients, who were classified by the American Society of Anaesthesiologists (ASA) as ASA I and II
2. Patients with the age of 18 and over
3. Patients who were diagnosed as in need of non-surgical orthograde root canal treatment of an asymptomatic tooth
4. Tooth without signs of previously initiated Root Canal Therapy

Exclusion Criteria:

1. Pregnant and lactating females
2. Patients with chronic periodontal diseases
3. Patients with sensitivity or adverse reactions to any medication or materials that were used throughout the treatment procedure
4. Patients with acute periapical periodontitis
5. Patients with acute periodontal abscess
6. Patients who could not abide by the follow-up time
7. Patients who used analgesics 1-week prior or antibiotics 1-month prior to treatment
8. Uncooperative patients
9. Teeth that cannot be made functional nor restored or difficult to access teeth with no importance (wisdom teeth)
10. Teeth with poor prognosis, for example, due to deep root caries or big root resorption
11. Teeth with more than/or equal 4 mm periodontal pocket depth
12. Teeth with an inaccessible root end
13. Teeth with apical resorption or a radiologically not clearly defined apex
14. Fractured teeth
15. Teeth with immature or open apices
16. Teeth with root apices extending into the maxillary sinus
17. Teeth with external resorption communicating with the pulp

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tan Firat EYÜBOĞLU, DDS, MDS, Principal Investigator — İstanbul Medipol University, Department of Endodontics, İstanbul/Türkiye; Mutlu ÖZCAN, DDS, MDS, Study Director — İstanbul Medipol University, Istanbul Turkey
Locations (1):
- İstanbul Medipol Universitesi, Faculty of Dentistry, Department of Endodontics, Istanbul, Unkapanı, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 10 participants who met all inclusion criteria and no exclusion criteria were randomized at 1 site to treatment between May 10, 2022 and May 31, 2022.
Pre-assignment Details: Subjects were randomized 1:1 on Study Day 0 to receive treatment either by manual irrigation with sodium hypochlorite NaOCl or by inertial cavitation-generating device.
Period: Overall Study
Arm/Group | Conventional Irrigation | Inertial Cavitation
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 5 participants baseline analysis was done in the conventional irrigation group and 5 participants baseline analysis was done in the inertial cavitation group. Overall 10 participants baseline analysis was conducted.
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Irrigation | Inertial Cavitation | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Customized [Mean (Standard Deviation); unit: years] — 10 participants were randomized to conventional irrigation or inertial cavitation groups and all 10 participants completed the study protocol.
  years
    Mean age of participants | 29.8 (13.8) | 26.8 (6.61) | 28.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 3 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Clinical Postoperative Pain
Description: Pain intensity levels were graded using Visual Analog Scale (VAS). This scale is a horizontal 100 mm bar, marked in every 10mm with two ends. One end (0) indicated "no pain" and the other end (100) indicated "worst pain possible". Categorization of pain scores is as follows: 0-4 mm = No Pain, 5-44 mm = Mild Pain, 45-74 mm = Moderate Pain, 75-100 mm = severe pain.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Irrigation | Inertial Cavitation
Number analyzed (Participants) | 5 | 5
score on a scale | 30.5 (10.6) | 20.6 (21.25)

2. Primary Outcome: Clinical Postoperative Pain
Description: as for outcome 1
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Irrigation | Inertial Cavitation
Number analyzed (Participants) | 5 | 5
score on a scale | 15.7 (8.36) | 21.2 (18.6)

3. Primary Outcome: Clinical Postoperative Pain
Description: as for outcome 1
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Irrigation | Inertial Cavitation
Number analyzed (Participants) | 5 | 5
score on a scale | 10.94 (8.82) | 12 (16.43)

4. Primary Outcome: Clinical Postoperative Pain
Description: as for outcome 1
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Irrigation | Inertial Cavitation
Number analyzed (Participants) | 5 | 5
score on a scale | 10.4 (10.32) | 12 (16.43)

5. Primary Outcome: Clinical Postoperative Pain
Description: as for outcome 1
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Irrigation | Inertial Cavitation
Number analyzed (Participants) | 5 | 5
score on a scale | 11.58 (16.2) | 4 (8.94)

ADVERSE EVENTS:
Time Frame: 1 week after treatment
Description: Endoclean Group (N=5) Control Group (N=5) Total (N=10) Completed 1w visit 5 5 10 Adverse device effect 0 0 0 Serious adverse device effect 0 0 0
Arm/Group | Conventional Irrigation | Inertial Cavitation
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT05374434/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT05374434/SAP_001.pdf